CLINICAL TRIAL: NCT05314296
Title: Multicenter Non-interventional Study of Osimertinib Administration in Patients With NSCLC Progression Occurred During or After Therapy With EGFR Tyrosine Kinase Inhibitors, With Confirmed Т790М Positive Mutation in EGFR Gene
Brief Title: Osimertinib for Russian EGFR T790M Mutation-positive NSCLC Patients Who Progressed on or After EGFR TKI Therapy
Acronym: TRUST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: N.N. Blokhin National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-17-13290
Record Dates: First submitted 2022-03-05; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-12

CONDITIONS: Non Small Cell Lung Cancer; T790M; EGFR Gene Mutation
Keywords: Tyrosine kinase inhibitor; Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess safety of Osimertinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with progression during or after therapy with a prior EGFR tyrosine kinase inhibitor (TKI), with confirmed Т790М positive mutation in EGFR gene.

DETAILED DESCRIPTION:
This study is a multicenter non-interventional retro- and prospective study of safety and efficacy of the Osimertinib administration in frames of Early Access Program (EAP) and real clinical practice in patients with locally advanced or metastatic non-small cell lung cancer that progressed during or after therapy with an EGFR tyrosine kinase inhibitor, with confirmed Т790М positive mutation in EGFR gene with explorative analysis of the set of mutations detected in plasma ctDNA taken after the progression on Osimertinib.

It is planned to include in the study approximately 70 patients in the Russian Federation (RF) who are participating or having completed their participation in EAP, or patients, who were treated with Osimertinib in real clinical practice.

For the patients participating in EAP and patients taking Osimertinib in real clinical practice, prospective data collection is planned after signing the informed consent form(ICF) for participation in the study. Data from those patients who completed participation in EAP or completed therapy with Osimertinib in real clinical practice will be gathered retrospectively, following the procedure of signing the ICF, or without it, if the procedure is not applicable (patient's death prior to the data collection).

Patients who are participating in EAP at the moment of inclusion into the TRUST study will receive therapy by Osimertinib at a dose of 80 mg a day orally, as a single dose. Patients will be treated according to the SmPC and local clinical regulations. Assessment of response to the therapy will be performed in accordance with RECIST 1.1.

From all patients included into the study will be performed retro- or prospective data collection of two-year-course of the disease starting from the time of first dose of Osimertinib.

For patients with progression of the disease on Osimertinib will be performed molecular-genetic testing of their plasma ctDNA at the time when the fact of the progression is registered.

During the study, each patient, for whom data will be collected prospectively, will undergo two data collection points: the first point (for signing of ICF and evaluation of eligibility criteria) and the final point, which will take place 2 years after the first dose of Osimertinib or at the time when therapy by Osimertinib is discontinued. Patients, for whom data will be collected retrospective, should underdo only the first visit for signing the ICF.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Osimertinib EAP and /or taking / completion therapy with Osimertinib in real clinical practice;
* Confirmed diagnosis of IIIB (locally advanced) or IV (metastatic) stages of NSCLC with T790M EGFRm;
* Progression of the disease that occurred during or after the therapy with first- or second-generation EGFR TKI

Exclusion Criteria:

* Participation in any other clinical study;
* Absence of data essential for obtaining all necessary information in full.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to include all the patients enrolled in an Osimertinib Early Access Program in Russia With Locally Advanced/Metastatic EGFR T790M Mutation-positive NSCLC and Prior Exposure to and progression on or after other EGFR TKI Therapy (presumably 45 to 50 subjects) and patients, who were treated with osimertinib in local clinical practice (presumably 20 to 25 subjects).
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one adverse event | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  By line of treatment:
  1. First line therapy
  2. Second line of therapy
  By treatment duration:
  1. Up to a year
  2. More than a year
  By effectiveness of therapy:
  1. Progression
  2. Stabilization
  3. Negative feedback
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21
Proportion of patients who discontinued therapy with Osimertinib | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  By line of treatment:
  1. First line therapy
  2. Second line of therapy
  By treatment duration:
  1. Up to a year
  2. More than a year
  By effectiveness of therapy:
  1. Progression
  2. Stabilization
  3. Negative feedback
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21

SECONDARY OUTCOMES:
Disease Control Rate and Objective Response Rate | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21
Progression-free survival | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21
Overall Survival | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21
Time to Treatment Discontinuation | Through study completion, an average of 5 years
  By sex:
  1. Male
  2. Female
  Previous targeted therapy:
  1. Yes
  2. No
  Variant of mutation:
  1. Exon 19
  2. Exon 21

OTHER OUTCOMES:
Exploratory outcome | Through study completion, an average of 5 years
  Percentage of patients who had been treated with other therapies prior to the start of therapy with Osimertinib.
  Percentage of patients who previously underwent targeted therapy and other types of therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution National Medical Research Center of Oncology named after N.N. N.N. Blokhin" of the Ministry of Health of Russia, Moscow, Russia